CLINICAL TRIAL: NCT00189384
Title: Randomized Controlled Trial of Intramuscular Ceftriaxone Versus Procaine Penicillin Versus Cotrimoxazole and Gentamicin for Management of Serious Bacterial Infections in Young Infants in Community Settings
Brief Title: Efficacy Study of Community-Based Treatment of Serious Bacterial Infections in Young Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC/SNL 11150-0902-50001-269
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Bacterial Infection; Sepsis; Infant, Newborn
Keywords: Neonatal sepsis; Neonatal pneumonia; Bacterial infections; Young infants; Neonate; Community; Developing country
MeSH Terms: conditions — Bacterial Infections; Sepsis; Neonatal Sepsis | interventions — Ceftriaxone; Penicillin G Procaine; Gentamicins; Trimethoprim, Sulfamethoxazole Drug Combination

INTERVENTIONS:
Drug: ceftriaxone, procaine penicillin and gentamicin, oral cotrimoxazole and gentamicin

SUMMARY:
Approximately one-third of neonatal deaths in developing countries are due to infections acquired through the birth canal and/or exposure to an unclean environment soon after birth. Current World Health Organization recommendations for the management of infants younger than 2 months of age who have serious bacterial infections involve hospitalization and parenteral therapy for at least 10 days with antibiotic regimens containing penicillin or ampicillin combined with an aminoglycoside.However, in many settings throughout the developing world, this is not currently possible, nor is this standard of care likely to be feasible in the near future. Several studies have reported that for a variety of sociocultural reasons many families are unable or unwilling to access hospital-based care and their sick young infants do not get hospitalized, and instead, receive a variety of home-based antibiotic therapies, or none at all. In our community field sites, approximately 70% of families refuse hospital referral for a sick newborn, despite provision of transport.

Thus, there is an urgent need to define the role of community/first-level facility-based care versus hospitalization for the management of young infants with serious bacterial infections, and the potential for community-based parenteral antibiotics as an alternative strategy in resource poor areas with high neonatal mortality rates. Bang and colleagues have demonstrated significant reductions in neonatal mortality from infections in an underdeveloped rural district in Maharashtra, India by a field-based case management approach which used oral cotrimoxazole and intramuscular gentamicin given for 7 days as treatment for neonates with sepsis.

This study is an equivalence randomized controlled trial (RCT) comparing once daily IM ceftriaxone injection to once daily IM procaine penicillin and gentamicin injection, to once daily intramuscular gentamicin injection and twice daily oral cotrimoxazole, given for 7 days in babies with clinically-diagnosed possible serious bacterial infection (pneumonia, or sepsis with or without local infections such as skin or umbilical infections) whose families refused referral to a hospital. After supplementary informed consent, patients meeting specific inclusion and exclusion criteria are randomly allocated to one of the three regimens being tested. The study hypothesis is that all 3 regimens will perform equally well in the treatment of sepsis in a first-level facility setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-59 days presenting to Young Infant community study site
* Clinical diagnosis of possible serious bacterial infection by study physician according to specified clinical criteria
* Parents refuse to accept referral care and sign (or thumb imprint) document stating this.
* Parents consent to community centre-based intramuscular antibiotic injections

Exclusion Criteria:

* Age over 59 days
* Presence of severe jaundice diagnosed clinically or by laboratory investigation (bilirubin > 12 g/dl in term and > 7 in pre-term baby).
* Presence of obvious meningitis (bulging fontanelle, observed seizures)
* Patient previously enrolled in antibiotic therapy trial
* Parents accept hospital referral
* Parents do not consent to any injectable therapy

Ages: 0 Years to 59 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 426
Dates: Start 2003-11; Study Completion 2005-12

PRIMARY OUTCOMES:
The primary outcome of success rate will be defined as patient cured or improved with the regimen assigned to, on day 7 of therapy.

SECONDARY OUTCOMES:
Completion rates
Adverse events
Relapse rates

CONTACTS AND LOCATIONS:
Overall Officials: Anita KM Zaidi, MBBS, SM, Principal Investigator — Department of Pediatrics, Aga Khan University
Locations (1):
- Aga Khan University community field sites, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Bang AT, Bang RA, Baitule SB, Reddy MH, Deshmukh MD. Effect of home-based neonatal care and management of sepsis on neonatal mortality: field trial in rural India. Lancet. 1999 Dec 4;354(9194):1955-61. doi: 10.1016/S0140-6736(99)03046-9. PMID 10622298
- [Background] Bang AT, Reddy HM, Deshmukh MD, Baitule SB, Bang RA. Neonatal and infant mortality in the ten years (1993 to 2003) of the Gadchiroli field trial: effect of home-based neonatal care. J Perinatol. 2005 Mar;25 Suppl 1:S92-107. doi: 10.1038/sj.jp.7211277. PMID 15791283
- [Background] Bang AT, Bang RA, Stoll BJ, Baitule SB, Reddy HM, Deshmukh MD. Is home-based diagnosis and treatment of neonatal sepsis feasible and effective? Seven years of intervention in the Gadchiroli field trial (1996 to 2003). J Perinatol. 2005 Mar;25 Suppl 1:S62-71. doi: 10.1038/sj.jp.7211273. PMID 15791280